CLINICAL TRIAL: NCT06045156
Title: Early Tirofiban Administration After Intravenous Thrombolysis in Acute Ischemic Stroke: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Early Tirofiban Administration After Intravenous Thrombolysis in Acute Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADVENT
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; intravenous thrombolysis; tirofiban
MeSH Terms: conditions — Ischemic Stroke | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban group (Active Comparator): Tirofiban infused with 0.4μg/kg/min for 30min and 0.1μg/kg/min until 24h after IVT
  Interventions: Drug: Tirofiban
- Tirofiban simulant group (Placebo Comparator): Tirofiban simulant infused with 0.4μg/kg/min for 30min and 0.1μg/kg/min until 24h after IVT
  Interventions: Drug: Tirofiban simulant

INTERVENTIONS:
Drug: Tirofiban — Tirofiban is a selective glycoproteinⅡb/Ⅲa receptor inhibitor, which inhibits platelet aggregation and thrombi formation
  Arms: Tirofiban group
Drug: Tirofiban simulant — Tirofiban simulant is placebo packed the same style as tirofiban
  Arms: Tirofiban simulant group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of early tirofiban administration in patients undergoing IVT

DETAILED DESCRIPTION:
Nearly half of acute ischemic stroke patients underwent intravenous thrombolysis (IVT) failed to achieve excellent functional outcome. Some studies reported that early administrated tirofiban, a selective glycoproteinⅡb/Ⅲa receptor inhibitor, may greatly improve the outcome of patients who received IVT, however they only recruited small sample size.

Thus, the investigators design early tirofiban administration after intravenous thrombolysis in acute ischemic stroke (ADVENT) trial, aiming to evaluate the efficacy and safety of early tirofiban administration in patients undergoing IVT.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years old;
2. Clinically diagnosed as acute ischemic stroke and received standard dose (0.25mg/kg) of tenecteplase IVT within 4.5 hours of onset;
3. Total National Institute of Health stroke scale (NIHSS)≥4 or single limb motor item score≥2, and total NIHSS≤15 after IVT;
4. Tirofiban or placebo treatment can be initiated within 6h after IVT;
5. mRS score before onset≤ 1;
6. Intracranial hemorrhage is ruled out by CT head after IVT;

Exclusion Criteria:

1. Received or plan to undergo bridge therapy;
2. Large area of infarct indicated by radiological imaging(≥1/3 of middle cerebral artery supply area);
3. Atrial fibrillation or suspected cardiac embolism;
4. Accompanied by epileptic seizures;
5. Using antiplatelet, anticoagulant or fibrinolytic agents within 24h before recruitment;
6. Active bleeding or tendency to bleed after receipt of intravenous thrombolysis;
7. Digestive system bleeding, urinary system bleeding, hemorrhagic retinopathy or other systemic bleeding events within 1 year;
8. Severe renal or liver insufficiency; ALT or AST>3 times of the upper limit of normal value or above; creatinine clearance rate<30 mL/min, creatinine>200μmol/L；
9. Life expectancy less than 3 months;
10. Pregnant or lactating women;
11. Known allergy to tirofiban;
12. Being enrolled or having been enrolled in other clinical trial within 3 months prior to this clinical trial.;
13. Patients who are unwilling to be followed up or likely to have poor treatment compliance;
14. Other situations that the researcher deems unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1084 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients of modified Rankin Scale (mRS)≤1 | 90±7 days
  mRS depicts functional outcome of stroke, which ranges from 0-6, mRS 0-1 represents excellent functional outcome

SECONDARY OUTCOMES:
Proportion of patients of mRS≤2 | 90±7 days
  mRS depicts functional outcome of stroke, which ranges from 0-6, mRS 0-2 represents favorable functional outcome
Distribution of mRS | 90±7 days
  mRS depicts functional outcome of stroke, which ranges from 0-6
National Institute of Health stroke scale (NIHSS) | 24 hours after IVT, 7 days
  National Institute of Health stroke scale (NIHSS) ranges from 0 to 42, a low value represents a better outcome

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage | within 24 hours of completion of study drug infusion, hospitalization
  Symptomatic intracranial hemorrhage is defined according to the ECASS Classification
Hemorrhagic transformation | 24 hours after IVT, hospitalization
  defined according to the ECASS Classification

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Guo ZN, Zhang KJ, Zhang P, Qu Y, Abuduxukuer R, Nguyen TN, Chen HS, Yang Y. Early tirofiban administration after intravenous thrombolysis in acute ischemic stroke (ADVENT): Study protocol of a multicenter, randomized, double-blind, placebo-controlled clinical trial. Eur Stroke J. 2024 Jun;9(2):510-514. doi: 10.1177/23969873231225069. Epub 2024 Jan 9. PMID 38196129